CLINICAL TRIAL: NCT03914924
Title: Effects of an Exercise and Lifestyle Education Program for People With Diabetes and Prediabetes: A Multicenter Randomized Controlled Trial
Brief Title: Effects of an Exercise and Lifestyle Education Program for People With Diabetes and Prediabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Collaborators: Federal University of Minas Gerais (Other); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Lilian Pinto da Silva, Professor, Principal Investigator, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DiabetesCollegeBrazil
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus; Prediabetes
Keywords: Diabetes Mellitus; Exercise; Health Education; Patient Education; Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Motor Activity; Health Education | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of two interventions: Exercise Program (Ex) or Exercise and Lifestyle Education Program (ExLE).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Program (Active Comparator): Ex: The participants will be submitted to only a 12-week exercise intervention.
  Interventions: Behavioral: Exercise Program
- Exercise and Lifestyle Education Program (Experimental): ExLE: The participants will be submitted to a 12-week intervention consisting of exercise and education.
  Interventions: Behavioral: Exercise Program; Behavioral: Lifestyle Education Program

INTERVENTIONS:
Behavioral: Exercise Program — On-site delivery: The supervised exercise sessions will be offered twice a week from the first to fourth weeks and once a week from the fifth week onwards. Each session lasts approximately 60 minutes.
  Remote delivery: The participants will attend an initial supervised exercise session delivered on-site. After this session, they will receive the exercise intervention through a website specific to the Ex program. Participants will receive weekly WhatsApp messages to remind them about the exercise routine.
  Independent of the delivery format all participants will receive counseling to accumulate at least 150 min of aerobic exercise per week.
Behavioral: Lifestyle Education Program — On-site delivery: The supervised exercise sessions will be offered twice a week from the first to fourth weeks and once a week from the fifth week onwards. Each session will last approximately 60 minutes. Participants will receive a printed version of the Diabetes College Guide containing twenty chapters and they will attend eighteen thirty-minute education classes.
  Remote delivery: The participants will attend an initial supervised exercise session delivered on-site. After this session, they will receive the interventions (exercise and education) through a website specific to the ExLE program. Participants will receive a printed version of the Diabetes College Guide, as well as, guidance on accessing the educational content on the website and weekly WhatsApp messages with reminders about educational content scheduled for that week.
  Independent of the delivery format all participants will receive counseling to accumulate at least 150 min of aerobic exercise per week.
  Arms: Exercise and Lifestyle Education Program

SUMMARY:
The purpose of this trial is to pragmatically investigate whether participation of people with diabetes and prediabetes in an Exercise and Lifestyle Education Program (i.e., exercise and education classes) results in better functional capacity, disease-related knowledge and behavior, and cardiometabolic health parameters when compared to Exercise Program (i.e., exercise class only). In addition, the effects of these interventions will be evaluated on other outcomes: program adherence, satisfaction with the program, quality of life, diet quality, depression, and morbidity associated with diabetes in the 6-month follow-up.

DETAILED DESCRIPTION:
The design is a multicenter, double-blind (outcomes assessors and data analysts), randomized and controlled trial with 2 parallel arms: Exercise Program (Ex) and Exercise and Lifestyle Education Program (ExLE). The sample size was calculated considering the ISWT distance as the primary outcome and based on a previous study that tested the effects of a comprehensive cardiac rehabilitation program on the same primary outcome in coronary patients. The calculation was made using R Software version 3.4.3 and considering the following parameters: moderate effect size (d = 0.20), the statistical power of 80%, an alpha level of 5%, a one-sided test, two arms, and three measurements. A total of 200 participants (100 per program) was required. Assuming a 20% attrition rate based on previous studies using educational intervention in Cardiac Rehabilitation patients, it will take 120 participants in each program to sign the consent form to have 200 participants complete the study.

Adults with diabetes and prediabetes will be recruited from public and private health services in two Brazilian cities (Belo Horizonte and Juiz de Fora). Volunteers will be allocated to participate in the program to which they were randomized and be invited for follow-up and reassessment after 6 months of program completion. In this sense, three assessments will be performed: pre-intervention (baseline), post-intervention, and 6 months post-program completion.

The baseline assessment will comprise an interview to obtain their clinical characteristics and sociodemographic data, medical history, vital signs measurement, electrocardiographic monitoring, and measurement of primary, secondary, and tertiary outcomes (other pre-specified outcome measures) through questionnaires and specific tests.

The number of patients approached, the date, and the reasons for inclusion/exclusion will be registered. With informed written consent from the patient, potentially eligible participants will be scheduled to come on-site to complete the baseline assessment. Eligible participants will be randomized to one of the 2 programs (Ex or ExLE). The generation of the randomized allocation sequence will be performed by the project coordinator using the software available on the website www.randomization.com. To ensure allocation concealment, the local research coordinators have the allocation sequence in a password-protected file. They will only provide randomization information to the research team member once it is confirmed the participant is eligible. Due to the nature of the intervention, participants and the research team members cannot be blind to the treatment allocated. However, an independent research member blinded to the group allocation will perform database management and analyses.

The programs (Ex and ExLE) will be delivered on-site or remotely based on internet access and technology literacy screening. Participants who attend these two conditions can choose the delivery format by which they would like to receive the program interventions. For those with no internet access and/or technology literacy, the delivery format of the program interventions will be on-site.

The 12-week exercise intervention consists of at least 150 min of aerobic exercise per week and 2 to 3 muscle-strengthening sessions per week from the 4th week of the intervention. The exercise sessions were structured in exercise sessions (on-site delivery) or exercise plans (remote delivery) as follows: warm-up (stretching exercises and slow walking), aerobic exercise (moderate-to-vigorous intensity walking according to the Borg rating of perceived exertion exercise scale modified), muscle-strengthening exercises (localized muscle endurance exercises that encompass the major muscle groups) and cool down (slow walking and stretching exercises). In the on-site delivery, participants will attend eighteen supervised exercise sessions and receive counseling for unsupervised physical exercise to accumulate at least 150 min/week. They should record their weekly exercise routine in an exercise diary. In the remote delivery, participants will access weekly exercise plans on the Ex program website, and only this program's participants will have access to this website link. They will also receive weekly follow-up text messages via WhatsApp with standardized reminders about exercise goals and the importance of keeping track of their exercise and reporting the exercise sessions in the exercise diary.

In addition to the exercise intervention, participants randomized to the ExLE program will receive a 12-week educational intervention developed based on the Diabetes CollegeTM curriculum (https://www.diabetescollege.ca), translated and culturally adapted for Brazilians living with diabetes and prediabetes. In the on-site delivery, participants will attend eighteen education classes based on the five pillars of Diabetes CollegeTM (treat diabetes, get active, eat healthy, feel well, and take control) and receive a printed version of the Patient Guide (A Guide to Help You Live and Thrive with Diabetes, containing 298 pages and 17 chapters organized into five sections). In the remote delivery, participants will access their weekly lesson plans on the ExLE program website, and only this program's participants will have access to this website link. The educational content consists of the following materials: (1) eighteen video lessons recorded by the research team based on the five pillars of Diabetes CollegeTM, lasting approximately 20 min; (2) twelve videos related to the topics of the week (THRiVE, i.e., videos that integrate principles of chronic disease management and behavior changes to help patients to develop self-management skills through goal setting and action planning); and (3) an printed version of the Patient Guide. In addition, as part of remote delivery, participants will receive weekly WhatsApp text messages from the research team to remind them about the materials in their lesson plan and the importance of keeping track of access to educational content and reporting it in the study diary.

All participants will be invited to the follow-up after the program's completion and the post-intervention assessment.

During the 6-month follow-up, participants will be instructed to record their Diabetes-related morbidity information on the standardized sheet developed by the research team. Research team members will make monthly phone calls to participants to remind them to perform this register properly. Besides that, to minimize dropouts to follow-up, the research team members will send email and phone reminders for patients about to come on-site to the 6-month follow-up assessment post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years old);
* Self-reported current history of prediabetes or Diabetes Mellitus (type 1 or type 2);
* No cognitive limitation (score ≥ 4 in the six-item screener);
* No vision limitations for reading;
* Literate;
* Written physician permission for exercising;
* No confirmed diagnosis of cardiovascular diseases such as unstable coronary artery disease (CAD), heart failure; use of a pacemaker and/or implantable cardioverter-defibrillator (ICD), intermittent claudication; no recent cardiovascular event or cardiac surgery (≤ 6 months);
* Participants not currently enrolled in a structured physical exercise program that follows diabetes guidelines.

Exclusion Criteria:

* Clinical decompensation that contraindicates the performance of physical exercises;
* Physical and/or mental limitations that will prevent the participant from physically exercising and/or understanding educational content;
* Complex ventricular arrhythmias (i.e., atrial flutter or atrial fibrillation, multiple atrial or ventricular ectopy, and atrioventricular or ventricular block).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Functional capacity | Change from Baseline Functional Capacity at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  This outcome will be measured by the Incremental Shuttle Walk Test (ISWT) distance.
Disease-related knowledge | Change from Baseline Disease-related knowledge at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment).
  This outcome will be assessed from the total score of the Brazilian Portuguese version of the DiAbeTes Education Questionnaire (DATE-Q). This questionnaire is a 20-item self-administered tool (answer options are: true or false or do not know) equally distributed in five domains (self-management, long-term complications, being active, healthy eating, and psychosocial well-being) based on the Diabetes College. The total score ranges from 0 to 20, and higher scores indicate better disease-related knowledge.

SECONDARY OUTCOMES:
Health Behavior: health literacy | Change from Baseline health literacy at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  This outcome will be measured by the Newest Vital Sign (NVS) tool score. This is a six-item toll regarding the information found on an accompanying nutrition label. Each correct response is worth one point with a total of six points possible. Scores equal or greater than four are evidence of adequate health literacy whereas scores below four are evidence of inadequate health literacy.
Health Behavior: physical activity level | Change from Baseline physical activity at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  This outcome will be measured from the total number of steps recorded by a pedometer during consecutive 7 days. For analysis of this outcome, the total number of steps recorded will be divided for seven in order to obtain the average number of steps/day for each participant. The level of physical activity will be classified from the average of steps/day, as follow: sedentary (<5000 steps/day); low active (5000-7499 steps/day); somewhat active (7500-9999 steps/day); active (≥10 000 steps/day) and highly active (>12 500 steps/day).
Health Behavior: exercise self-efficacy | Change from Baseline Exercise Self-efficacy at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  This outcome will be assessed from the total score of the Brazilian Portuguese version of Bandura's exercise self-efficacy scale. This is an 18-item self-administered tool which item contents are related to situations that may compromise the adherence to regular physical exercising, e. g. when feeling tired or during the holidays. The respondent should indicate from 0 (no confident) to 100 (very confident) how much confidence he or she has about maintaining the physical exercise routine face of the situation described in that item. The total score is the average from the eighteen items scores, and higher total scores indicate great exercise self-efficacy.
Health Behavior: adherence to standard Mediterranean food elements | Change from baseline adherence to standard Mediterranean food elements at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  This outcome will be assessed from the total score of the Brazilian Portuguese version of the Mediterranean diet scale (MDS). The MDS has 13 items which quantitatively assess adherence to standard Mediterranean food elements [21]. The answer options are dichotomous: yes and no. Some questions have pictures and examples to help participants to answer the questions. One point is scored for each yes answered. Total scores range from 0 to 13. Scores below 5 indicate poor adherence to the MedDiet, and scores greater than 10 indicate high adherence.
Health Behavior: medication adherence | Change from Baseline Medication adherence at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  This outcome will be assessed from the total score of the Brazilian version of the Measure of Adherence to Oral Antidiabetic and Insulin Treatments questionnaire (MAT ADOs and MAT insulin), consisting of 7 items. The total score is determined by the average of scores obtained for each item.Higher scores mean more adherence.
Cardiometabolic Health Parameter: glycemic control | Change from Baseline blood sugar level at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  This outcome will be assessed from the glycated hemoglobin (A1c) level obtained in routine tests dated no more than three months before the study assessment point.
Cardiometabolic Health Parameter: anthropometric characteristics | Change from Baseline BMI and waist circumference at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  This outcome will be measured by the body mass index (BMI - kg/m2) and the waist circumference.
Cardiometabolic Health Parameter: cardiac autonomic control | Change from Baseline Cardiac autonomic control at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  This outcome will be assessed from heart rate variability (HRV) indexes.

OTHER OUTCOMES:
Program adherence | 12 weeks (post-intervention assessment).
  This outcome will be measured by the attendance rate in the program for each participant.
Satisfaction with the program | 12 weeks (post-intervention assessment).
  This outcome will be measured by questionnaires developed by the researchers. A questionnaire will assess the satisfaction with the exercise program and will be responded to by participants from the two programs (ExLE and Ex). Other one will assess the satisfaction with the learning tools of Diabetes College and will be responded to only by participants of the Exercise and Lifestyle Education Program (ExLE).
Quality of life level | Change from Baseline Quality of life at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  Quality of life level will be evaluated using the the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36). This questionnaire assesses 8 physical and mental health domains: Physical Functioning, Social Functioning, Role-Physical, Bodily Pain, Mental Health, Role-Emotional,Vitality and General Health. For each domain, item scores are coded, summed, and transformed, with final values (expressed as a percentage) ranging from 0 (worst health) to 100 (best health).
Depression | Change from baseline depression at 12 weeks (post-intervention assessment) and 6 months (follow-up assessment)
  This outcome will be measured by the Brazilian version of the Center for Epidemiological Scale - Depression (CESD). This is a 20-item tool used to rate how often the interviewed experienced symptoms associated with depression over the past week, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = rarely or none of the time, 1 = some or little of the time, 2 = moderately or much of the time, 3 = most or almost all the time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Diet quality | Change from baseline diet quality at 6 months (follow-up assessment)
  This outcome will be measured by a quantitative food frequency questionnaire (FFQ) at baseline (pre-intervention assessment) and 6 months post-intervention (follow-up assessment) and by a qualitative FFQ at the end of 12-week intervention (post-intervention assessment). The quantitative FFD that will be used contains 104 items distributed in eight food groups ("cereals, tubers, roots, and derivatives"; "vegetables and legumes"; "fruits"; "beans"; "meat and eggs"; "milk and dairy products"; "oils and fats," and "sugars and sweets"), as well as 11 items investigating beverages, 4 items investigating oilseeds and 1 item investigating food supplement.
Morbidity associated with diabetes | 6 months after post-intervention assessment (follow-up assessment).
  This outcome will be assessed through the participant's record during the 6-month follow-up regarding the following parameters: number of hospitalizations associated with diabetes, the occurrence of acute complications and diagnoses of chronic complications of diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Lilian P da Silva, PhD, Principal Investigator — University Federal of Juiz de Fora
Locations (2):
- Brazil (2):
  - Federal University of Minas Gerais, Belo Horizonte, Minas Gerais
  - Federal University of Juiz de Fora, Juiz de Fora, Minas Gerais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Introduction: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S1-S2. doi: 10.2337/dc18-Sint01. No abstract available. PMID 29222369
- [Background] Sociedade Brasileira de Diabetes. 2017. "Diretrizes Da Sociedade Brasileira de Diabetes 2017-2018." (D): 257-63.
- [Result] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Result] Fiocco AJ, Scarcello S, Marzolini S, Chan A, Oh P, Proulx G, Greenwood C. The effects of an exercise and lifestyle intervention program on cardiovascular, metabolic factors and cognitive performance in middle-aged adults with type II diabetes: a pilot study. Can J Diabetes. 2013 Aug;37(4):214-219. doi: 10.1016/j.jcjd.2013.03.369. Epub 2013 Aug 2. PMID 24070883
- [Result] Kuziemski K, Slominski W, Jassem E. Impact of diabetes mellitus on functional exercise capacity and pulmonary functions in patients with diabetes and healthy persons. BMC Endocr Disord. 2019 Jan 3;19(1):2. doi: 10.1186/s12902-018-0328-1. PMID 30606177
- [Result] Odgers-Jewell K, Ball LE, Kelly JT, Isenring EA, Reidlinger DP, Thomas R. Effectiveness of group-based self-management education for individuals with Type 2 diabetes: a systematic review with meta-analyses and meta-regression. Diabet Med. 2017 Aug;34(8):1027-1039. doi: 10.1111/dme.13340. Epub 2017 Mar 20. PMID 28226200
- [Result] Chaves GSDS, Ghisi GLM, Grace SL, Oh P, Ribeiro AL, Britto RR. Effects of comprehensive cardiac rehabilitation on functional capacity in a middle-income country: a randomised controlled trial. Heart. 2019 Mar;105(5):406-413. doi: 10.1136/heartjnl-2018-313632. Epub 2018 Oct 3. PMID 30282639
- [Result] Machado CCDS, Malaguti C, Trevizan PF, Ezequiel DGA, Seixas MB, da Silva LP. Psychometric validation of the Brazilian Portuguese version of Bandura's exercise self-efficacy scale in diabetes patients. J Diabetes Metab Disord. 2020 Jul 15;19(2):925-932. doi: 10.1007/s40200-020-00581-6. eCollection 2020 Dec. PMID 33520812
- [Result] Felix CMM, Ghisi GLM, Seixas MB, Batalha APDB, Ezequiel DGA, Trevizan PF, Pereira DAG, Silva LPD. Translation, cross-cultural adaptation, and psychometric properties of the Brazilian Portuguese version of the DiAbeTes Education Questionnaire (DATE-Q). Braz J Phys Ther. 2021 Sep-Oct;25(5):583-592. doi: 10.1016/j.bjpt.2021.03.003. Epub 2021 Mar 26. PMID 33824060
- [Result] Teixeira RL, Jansen AK, Pereira DA, Ghisi GLM, Silva LPD, Cisneros LL, Britto RR. Brazilian Portuguese version of the Mediterranean diet scale: Translation procedures and measurement properties. Diabetes Metab Syndr. 2021 Jul-Aug;15(4):102165. doi: 10.1016/j.dsx.2021.06.002. Epub 2021 Jun 5. PMID 34186358
- [Result] Ghisi GLM, Seixas MB, Pereira DS, Cisneros LL, Ezequiel DGA, Aultman C, Sandison N, Oh P, da Silva LP. Patient education program for Brazilians living with diabetes and prediabetes: findings from a development study. BMC Public Health. 2021 Jun 26;21(1):1236. doi: 10.1186/s12889-021-11300-y. PMID 34174860
- [Result] Seixas MB, Pereira DAG, Ghisi GLM, Batalha APDB, Santos CVO, Ponciano IC, Oh P, Silva LPD. Exercise and Lifestyle Education program for Brazilians living with prediabetes and diabetes: A pilot randomized trial. Diabetes Metab Syndr. 2022 Oct;16(10):102614. doi: 10.1016/j.dsx.2022.102614. Epub 2022 Sep 6. PMID 36115088
- [Result] Seixas MB, Ghisi GLM, Oh P, Pereira DS, Moreira APB, Jansen AK, Batalha APDB, Candido GDN, Almeida JA, Pereira DAG, Silva LPD. Feasibility of Remote Delivering an Exercise and Lifestyle Education Program for Individuals Living with Prediabetes and Diabetes in Brazil. Int J Environ Res Public Health. 2022 Dec 12;19(24):16697. doi: 10.3390/ijerph192416697. PMID 36554577
- [Result] Boas LC, Lima ML, Pace AE. Adherence to treatment for diabetes mellitus: validation of instruments for oral antidiabetics and insulin. Rev Lat Am Enfermagem. 2014 Jan-Feb;22(1):11-8. doi: 10.1590/0104-1169.3155.2386. PMID 24553698
- [Derived] Silva LPD, Batalha APDB, Ghisi GLM, Seixas MB, Cisneros LL, Jansen AK, Moreira APB, Pereira DS, Britto RR, Pereira DAG, Trevizan PF, Oh P. Effects of an Exercise and Lifestyle Education Program in Brazilians living with prediabetes or diabetes: study protocol for a multicenter randomized controlled trial. Trials. 2024 Oct 21;25(1):701. doi: 10.1186/s13063-024-08535-6. PMID 39434107
- See also: Diabetes College — https://www.healtheuniversity.ca/EN/DiabetesCollege